CLINICAL TRIAL: NCT01765049
Title: Prospective Study Analyzing Value of Breast Density Change Predicting ENdocrine Therapy Response in Postmenopausal Women Taking Adjuvant ARomatase Inhibitor
Brief Title: Breast Density Change Predicting Response to Adjuvant Aromatase Inhibitor
Acronym: DEAR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SNUHBCC001
Record Dates: First submitted 2013-01-08; First posted 2013-01-10 (Estimated); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Invasive Breast Cancer; Estrogen Receptor Positive Breast Cancer
Keywords: breast density change; endocrine therapy response; aromatase inhibitor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Postoperatively collected specimen (normal and cancer tissue) Preoperatively collected blood sample
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Breast density change after short term use of aromatase inhibitor in postmenopausal ER positive breast cancer would predict endocrine responsiveness

DETAILED DESCRIPTION:
Inclusion criteria ER positive breast cancer Postmenopause women Older than 60yr S/P bilateral salphingo-oophorectomy No menstruation history within 1yr and FSH>30mIU/mL Ipsilateral invasive breast cancer Undergone curative resection No evidence of distant metastasis Capable of breast MRI

ELIGIBILITY:
Inclusion Criteria:

* ER positive invasive breast cancer Postmenopause women age 60yrs or older s/p bilateral salphingo-oophorectomy No history of menstruation and FSH>30mIU Planned for aromatase inhibitor Unilateral breast cancer Curative resection No evidence of distant metastasis

Exclusion Criteria:

* Bilateral breast cancer Male breast cancer Acceptable for breast MRI Pregnancy or lactation

Max Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Postmenopausal women with ER positive invasive breast cancer taking adjuvant endocrine therapy with aromatase inhibitor
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2013-01; Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 5 year
  recurrence locoregional distant metastasis Confirmed by clinical imaging or pathology

SECONDARY OUTCOMES:
breast density change | 6mos, 1yr, 2yr
  breast density change measured by cumulus(mammogram) and MRI(bilateral breast MRI) imagings taken after 6mos, 1yr, 2yr after endocrine therapy initiation

OTHER OUTCOMES:
overall survival | 5 year
  disease specific survival overall survival during 5yr follow up

CONTACTS AND LOCATIONS:
Overall Officials: Wonshik Han, MD PhD, Principal Investigator — SNUH
Locations (1):
- Seoul National University Hospital, Seoul, South Korea